CLINICAL TRIAL: NCT04068077
Title: Application of High Resolution Optical Coherence Tomography in Skin Disease: Amyloidosis and Differential Diagnosis
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-10-019A
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Amyloidosis
Keywords: optical coherence tomography (OCT); amyloidosis; pigmented diseases; skin diseases; dermatology; pathology; H&E stain
MeSH Terms: conditions — Amyloidosis; Skin Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients with amyloidosis and other indistinguishable diseases
  Interventions: Device: ApolloVue™ S100 image system, Viper1-S003

INTERVENTIONS:
Device: ApolloVue™ S100 image system, Viper1-S003 — The device is an in vivo non-invasive optical coherence tomography and will be used to obtain at least 6 medical images of normal and lesional skin, respectively, for experimental group.

SUMMARY:
Amyloidosis is caused by the misfolding protein accumulated in tissue, which affects the function of the organs. In addition to the primary cutaneous amyloidosis, a skin lesion may also appear in another classification - systemic amyloidosis. Physicians can confirm diagnosis of the above classification by skin biopsy.

Primary cutaneous amyloidosis is common in Asia and South America. In Taiwan, 80 people are diagnosed with primary cutaneous amyloidosis in every 100,000 people. Among the disease, macular amyloidosis and lichen amyloidosis are the most common subtypes. Primary cutaneous amyloidosis can cause severe itching, pigmentation, and skin keratosis, and further affect the social behavior of patients. The etiology of primary cutaneous amyloidosis is currently unclear, possibly due to genetic variations or viral infection. Typical primary cutaneous amyloidosis can be diagnosed by clinical manifestations, however, if the location or appearance of a lesion is atypical, the disease will be indistinguishable from other pigmented diseases, and further need a biopsy. If physicians can use a rapider and more accurate assistance tool to evaluate disease first, it will improve the accuracy of clinical diagnosis, relieve patient of suffering from biopsy, and further use medical resources more effectively.

Optical coherence tomography (OCT) is a kind of optical imaging medical system. It generates images by detecting the variations in refractive indexes of the various components in soft tissues. Apollo Medical Optics, Ltd. (AMO)'s OCT device (ApolloVue™ S100 image system, Viper1-S003) acquires real-time in vivo skin tissue tomograms with cellular resolution which provides a non-invasive, non-radioactive and rapid image acquisition.

In this study, AMO's OCT will be used to observe features in tomograms of primary cutaneous amyloidosis and that of other indistinguishable diseases, compare the correspondence of tomograms with pathological sections, induct features in tomograms specific to primary cutaneous amyloidosis and other indistinguishable diseases, and further establish an OCT database of primary cutaneous amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with suspected primary cutaneous amyloidosis and other indistinguishable diseases
* Patients with no open wounds

Exclusion Criteria:

* Patients with a transcutaneous infectious disease
* Patients under the age of 20
* Vulnerable populations, including: pregnant women, handicapped, and homelessness
* Patient cannot cooperate in examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from experimental group will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clear tissue characteristics of amyloidosis and/or other pigmented diseases in tomograms | 1 year
  Number of subjects with clear tissue characteristics of tomograms will be compared to that with unclear tissue characteristics to identify the effect of the OCT on scanning amyloidosis and other pigmented diseases at study completion.
Number of subjects with the distinction between skin lesion and normal skin in tomograms | 1 year
  Number of subjects with the distinction between skin lesion and normal skin in tomograms will be compared to that with no distinction to verify the specific diseases that can be distinguished from normal skin by the OCT at study completion.

SECONDARY OUTCOMES:
Number of subjects with the distinction between amyloidosis and other pigmented diseases in tomograms | 1 year
  Number of subjects with the distinction between amyloidosis and other pigmented diseases in tomograms will be compared to that with no distinction to verify the effect of the OCT on distinguishing amyloidosis from other pigmented diseases at study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Dar Lee, M.D., Ph. D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chuang YY, Lee DD, Lin CS, Chang YJ, Tanaka M, Chang YT, Liu HN. Characteristic dermoscopic features of primary cutaneous amyloidosis: a study of 35 cases. Br J Dermatol. 2012 Sep;167(3):548-54. doi: 10.1111/j.1365-2133.2012.11066.x. PMID 22632408
- [Background] Lei W, Ai-E X. Reflectance confocal microscopy for the characterization of primary cutaneous amyloidosis: a pilot study. Skin Res Technol. 2017 Aug;23(3):441-443. doi: 10.1111/srt.12343. Epub 2017 Jan 12. No abstract available. PMID 28083882
- [Background] Esmat SM, Fawzi MM, Gawdat HI, Ali HS, Sayed SS. Efficacy of different modes of fractional CO2 laser in the treatment of primary cutaneous amyloidosis: A randomized clinical trial. Lasers Surg Med. 2015 Jul;47(5):388-95. doi: 10.1002/lsm.22361. Epub 2015 May 6. PMID 25946210
- [Background] Al Yahya RS. Treatment of primary cutaneous amyloidosis with laser: a review of the literature. Lasers Med Sci. 2016 Jul;31(5):1027-35. doi: 10.1007/s10103-016-1917-8. Epub 2016 Mar 16. PMID 26984345
- [Background] Chang CK, Tsai CC, Hsu WY, Chen JS, Liao YH, Sheen YS, Hong JB, Lin MY, Tjiu JW, Huang SL. Errata: Segmentation of nucleus and cytoplasm of a single cell in three-dimensional tomogram using optical coherence tomography. J Biomed Opt. 2017 Mar 1;22(3):39801. doi: 10.1117/1.JBO.22.3.039801. No abstract available. PMID 28300273
- [Background] Chiu YK, Chen WL, Tsai CT, Yang CH, and Huang SL. A high en-face resolution AS-OCT providing quantitative ability to measure layered corneal opacities. European Conferences on Biomedical Optics, Munich Germany, 25-29, 2017.
- [Background] Wang SC, Hsu CY, Yang TT, Jheng DY, Yang TI, Ho TS, Huang SL. Laser-diode pumped glass-clad Ti:sapphire crystal fiber laser. Opt Lett. 2016 Jul 15;41(14):3217-20. doi: 10.1364/OL.41.003217. PMID 27420499
- [Background] Wang SC, Yang TI, Jheng DY, Hsu CY, Yang TT, Ho TS, Huang SL. Broadband and high-brightness light source: glass-clad Ti:sapphire crystal fiber. Opt Lett. 2015 Dec 1;40(23):5594-7. doi: 10.1364/OL.40.005594. PMID 26625059
- [Background] Tsai CC, Chang CK, Hsu KY, Ho TS, Lin MY, Tjiu JW, Huang SL. Full-depth epidermis tomography using a Mirau-based full-field optical coherence tomography. Biomed Opt Express. 2014 Aug 8;5(9):3001-10. doi: 10.1364/BOE.5.003001. eCollection 2014 Sep 1. PMID 25401013
- [Background] Ho TS, Yeh P, Tsai CC, Hsu KY, Huang SL. Spectroscopic measurement of absorptive thin films by spectral-domain optical coherence tomography. Opt Express. 2014 Mar 10;22(5):5675-83. doi: 10.1364/OE.22.005675. PMID 24663908
- [Background] Cheng NC, Hsieh TH, Wang YT, Lai CC, Chang CK, Lin MY, Huang DW, Tjiu JW, Huang SL. Cell death detection by quantitative three-dimensional single-cell tomography. Biomed Opt Express. 2012 Sep 1;3(9):2111-20. doi: 10.1364/BOE.3.002111. Epub 2012 Aug 13. PMID 23024905